CLINICAL TRIAL: NCT01361139
Title: Detection and Characterization of Cardio-Pulmonary Patho-Physiological States and Diseases by Transthoracic Parametric Doppler (TPD)
Brief Title: Diagnosis of Cardio-Pulmonary Pathology Using Transthoracic Parametric Doppler (TPD)
Status: Completed | Type: Observational
Sponsor: Echosense Ltd. (Industry)
Collaborators: Clalit Health Services, Haifa and West Galilee (Other)
Responsible Party: Sponsor
Other Study IDs: DOP09
Record Dates: First submitted 2011-05-25; First posted 2011-05-26 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2012-06

CONDITIONS: Lung Disease, Chronic Obstructive; Lung Disease, Interstitial; Asthma; Sarcoidosis; Hypertension, Pulmonary
Keywords: Chronic obstructive lung disease; Interstitial lung disease; Asthma; Sarcoidosis; Pulmonary hypertension; Ultrasound; Doppler; Lung disease diagnosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Asthma; Sarcoidosis; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study that seeks to characterize data obtained from patients with a variety of lung diseases using ultrasound signals obtained from the lung tissue. A standard ultrasound instrument in the doppler mode (not the imaging mode used in examination of pregnant women for instance) is placed on the chest wall and the unique software the investigators have developed analyzes the signal reflected back from within the lung. On the basis of pilot studies performed previously the investigators expect to receive different signals from different diseases. The investigators seek to further characterize these signals to enable accurate diagnosis of different lung diseases using our technology.

ELIGIBILITY:
INCLUSION CRITERIA

Age 18 years or older Patients who are clinically suspected of having pulmonary, cardiac or Cardio-pulmonary disease preferably any one or more of the conditions listed below:

* Patients with CHF
* Patients with pulmonary hypertension with documented right heart catheterization data
* Patients with COPD in two subgroups:

  * Emphysema, (evidence of emphysema on High Resolution Computed Tomography, (HRCT) and airflow limitation of GOLD II severity who have had Carbon Monoxide Diffusing capacity, (DLCO) and Residual Volume(RV) measured, or patients without HRCT with measurements of lung volumes and diffusing capacity with Total Lung Capacity (TLC) ≥1.0 predicted, RV/TLC ≥0.4, DLCO ≤ 0.7 predicted.
  * Chronic Bronchitis (No evidence of Emphysema on HRCT and/or no evidence of air-trapping or reduced DLCO.)
* Patients with asthma according to ATS/ERS definition,
* Patients with interstitial lung disease (ILD) of any etiology including sarcoidosis diagnosed by HRCT in sub groups as follows:

  * Mild ILD (TLC 0.71-0.79 predicted, DLCO ≥ 0.71 predicted)
  * Moderate and severe ILD (TLC ≤ 0.7 predicted, DLCO ≤ 0.7 predicted)
* Signed informed consent.
* Patients with sarcoidosis without evidence of parenchymal lung disease defined as normal DLCO and/or HRCT.

EXCLUSION CRITERIA

* Patients unable to cooperate.
* Inability to assume a semi-reclining or supine position
* Patients with severe chest wall deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to a large hospital-affiliated community lung clinic.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Diagnose specific pattern of the LDS signals as Power and Velocity in pulmonary diseases in comparison to controls. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiler, MD, Study Director — Echosense Ltd.; Uzi Milman, MD, Principal Investigator — Clalit Health Services
Locations (2):
- Israel (2):
  - Regional Pulmonary Clinic, Clalit Health Services, Haifa
  - Regional Clinic for Pulmonary Disease, Haifa and Western Galilee, Clalit Health Services, Haifa